CLINICAL TRIAL: NCT03295266
Title: An Open-Label Study to Investigate the Single-Dose Pharmacokinetics of MK-3866 When Administered to Subjects With Moderate and Severe Hepatic Impairment
Brief Title: Single-Dose Pharmacokinetics of MK-3866 in Participants With Hepatic Impairment (MK-3866-006)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business and program changes
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3866-006; MK-3866-006 (Other: Merck Protocol Number)
Record Dates: First submitted 2017-09-25; First posted 2017-09-27 (Actual); Results first posted 2019-11-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-10

CONDITIONS: Hepatic Insufficiency; Antibacterial Agents
MeSH Terms: conditions — Hepatic Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Moderate Hepatic Impairment (Panel A) (Experimental): Participants with moderate HI (estimated glomerular filtration rate [eGFR] of ≤60mL/min/1.73m^2) receive a single IV dose of MK-3866 (150 mg) on Day 1.
  Interventions: Drug: MK-3866
- Severe Hepatic Impairment (Panel B) (Experimental): Participants with severe HI (eGFR of ≤50 mL/min/1.73m^2) receive a single IV dose of MK-3866 (150 mg) on Day 1.
  Interventions: Drug: MK-3866
- Healthy Matched Controls (Panel C) (Experimental): Healthy participants receive a single IV dose of MK-3866 (150 mg) on Day 1.
  Interventions: Drug: MK-3866

INTERVENTIONS:
Drug: MK-3866 — Single IV infusion of MK-3866 150 mg administered over 30 minutes at Hour 0 on Day 1 of treatment period.

SUMMARY:
This is an open-label, single-dose, Phase 1 study to evaluate the pharmacokinetics (PK) of intravenous (IV) MK-3866 in participants with moderate and severe hepatic impairment (HI) compared to that of matched healthy participants. The primary purpose of this study is to understand the effect of HI on the plasma PK of MK-3866 in order to guide dosing recommendations for participants with HI. This study will also evaluate the safety and tolerability of MK-3866 in participants with moderate and severe HI.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index ≥19 & ≤40 kg/m^2
* Continuous non-smoker prior to screening & enrollment
* HI Participants: Baseline health judged to be stable based on medical history (except for the HI condition), physical examination, vital signs, electrocardiograms, & laboratory safety tests
* Healthy control participants: Is medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, or electrocardiograms
* HI Participants: Diagnosis of chronic (>6 months), stable (no acute episodes of illness within the previous 2 months due to deterioration in hepatic function) HI with features of cirrhosis
* HI Participants - Panel A (moderate HI) only: score on the Child-Pugh scale from 7 to 9 (moderate HI). At least 3 participants must have a score of 2 or higher on at least one of the laboratory parameters (i.e., albumin, international normalized ratio, and/or bilirubin) on the Child-Pugh scale
* HI Participants - Panel B (severe HI) only: Score on the Child-Pugh scale from 10 to 15 (severe HI)
* Is completely informed of the unknown risks of pregnancy & agrees not to become pregnant or father a child during time in study
* For a female of childbearing potential: is either sexually inactive (abstinent) for 14 days prior to dosing & throughout the study or is using an acceptable birth control method
* Non-vasectomized male: Participants must agree to use a condom with spermicide or abstain from sexual intercourse from dosing until 90 days after dosing

Exclusion Criteria:

* Mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study
* Has a history or presence of clinically significant medical or psychiatric condition or disease (other than HI - Panels A & B) that might confound the results of the study or poses an additional risk to the participant. Remote history of cholecystectomy that is not an active issue may be included.
* Panels A & B: Has a clinically significant history of cancer. Remote history with full cure or limited disease with complete resection (cure) may be included
* Has a history of drug/alcohol abuse within the past 6 months prior to dosing (Panels A & B) or within the past 2 years prior to dosing (Panel C [Healthy controls])
* Panels A & B: Consumes more than 3 glasses of alcoholic beverages (1 glass approximately equivalent to: beer [354 mL/12 ounces], wine [118 mL/4 ounces], or distilled spirits [29.5 mL/1 ounce]) per day, within 6 months of screening. Participants that consume 4 glasses of alcoholic beverages/day may be enrolled
* Panels A & B: Consumes excessive amounts, defined as more than 6 servings (1 serving approximately equivalent to 120 mg of caffeine), of coffee, tea, cola, energy-drinks, or other caffeinated beverages/day
* Panels A & B: Has a history of a liver transplant
* Has a history or presence of hypersensitivity or idiosyncratic reaction to the study drugs or related compounds
* Has moderate or severe renal insufficiency (estimated glomerular filtration rate of ≤60 mL/min/1.73 m2 for moderate HI or healthy control participants or ≤50 mL/min/1.73 m2 for severe HI participants)
* Panel C: Has positive macroscopic urine protein at screening (trace protein by dipstick allowed)
* Is a female participant who is pregnant or lactating
* Has positive results for the urine or breath alcohol screen and/or urine drug screen at screening
* Has positive results at screening for human immunodeficiency virus (HIV) (Panels A & B) or for HIV, HBsAg, or hepatitis C virus (HCV) (Panel C)
* Panels A & B: Participants with active HCV infection or hepatitis B virus (HBV) infection. Participants with prior/inactive HCV infection or past HBV infection may be enrolled.
* Is unable to refrain from or anticipates use of any medication or substance prohibited in study
* Has taken amiodarone at any time in their life

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (2):
- United States (2):
  - Clinical Pharmacology of Miami ( Site 0001), Hialeah, Florida
  - Orlando Clinical Research Center ( Site 0002), Orlando, Florida

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study terminated prior to enrollment of any healthy control participants.
Pre-assignment Details: Participants with moderate or severe hepatic impairment (HI) based on estimated glomerular filtration rate (eGFR) were enrolled at 2 study centers in the US.
Groups:
- Moderate Hepatic Impairment (Panel A): Participants with moderate HI (eGFR of ≤60mL/min/1.73m^2) received a single IV dose of MK-3866 (150 mg infused over 30 minutes) on Day 1.
- Severe Hepatic Impairment (Panel B): Participants with severe HI (eGFR of ≤50 mL/min/1.73m^2) received a single IV dose of MK-3866 (150 mg infused over 30 minutes) on Day 1.
Period: Overall Study
Arm/Group | Moderate Hepatic Impairment (Panel A) | Severe Hepatic Impairment (Panel B)
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderate Hepatic Impairment (Panel A) | Severe Hepatic Impairment (Panel B) | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.0 (5.96) | 56.0 (8.98) | 58.2 (7.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 4 | 3 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of MK-3866 From Time 0 to Infinity (AUC0-∞)
Description: AUC0-∞ is determined for the period up to 72 hours post-single dose. AUC0-∞ is an estimate of total plasma exposure from dosing to (extrapolated) infinity.
Time Frame: Predose, 0.5 (end of infusion), 0.75, 1, 1.5, 2, 3, 4.5, 6, 8, 10, 12, 24, 48, and 72 hours postdose
Population: All treated participants with data available are included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*µM
Arm/Group | Moderate Hepatic Impairment (Panel A) | Severe Hepatic Impairment (Panel B)
Number analyzed (Participants) | 5 | 4
hour*µM | 71.4 (7.3) | 58.6 (41.4)

2. Primary Outcome: Area Under the Concentration-time Curve of MK-3866 From Time 0 to Last Quantifiable Concentration (AUC0-last)
Description: AUC0-last is determined for the period up to 72 hours post-single dose. AUC0-last is an estimate of total plasma exposure from dosing to the time of last measurable sample.
Time Frame: Predose, 0.5 (end of infusion), 0.75, 1, 1.5, 2, 3, 4.5, 6, 8, 10, 12, 24, 48, and 72 hours postdose
Population: All treated participants with data available are included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*µM
Arm/Group | Moderate Hepatic Impairment (Panel A) | Severe Hepatic Impairment (Panel B)
Number analyzed (Participants) | 5 | 4
hour*µM | 70.7 (7.4) | 57.9 (42.2)

3. Primary Outcome: Area Under the Concentration-time Curve of MK-3866 From Time 0 to 24 Hours (AUC0-24hr)
Description: AUC0-24 is determined for the period up to 24 hours post-single dose. AUC0-24 is an estimate of total daily plasma exposure from dosing to 24 hours postdose.
Time Frame: Predose, 0.5 (end of infusion), 0.75, 1, 1.5, 2, 3, 4.5, 6, 8, 10, 12, and 24 hours postdose
Population: All treated participants with data available are included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*µM
Arm/Group | Moderate Hepatic Impairment (Panel A) | Severe Hepatic Impairment (Panel B)
Number analyzed (Participants) | 5 | 3
hour*µM | 67.6 (7.5) | 54.6 (34.5)

4. Primary Outcome: Concentration at the End of Infusion (Ceoi) of MK-3866
Description: The plasma sample collected at end-of-infusion (0.5 hours postdose) was used to determine Ceoi.
Time Frame: 0.5 (end of infusion) hours postdose
Population: All treated participants with data available are included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µM
Arm/Group | Moderate Hepatic Impairment (Panel A) | Severe Hepatic Impairment (Panel B)
Number analyzed (Participants) | 5 | 4
µM | 19.2 (22.0) | 11.0 (30.4)

5. Primary Outcome: Time to Maximum Concentration (Tmax) of MK-3866
Description: Tmax is the time at which the maximum plasma drug concentration is detected.
Time Frame: Predose, 0.5 (end of infusion), 0.75, 1, 1.5, 2, 3, 4.5, 6, 8, 10, 12, 24, 48, and 72 hours postdose
Population: All treated participants with data available are included.
Measure: Median (Full Range); unit: hours
Arm/Group | Moderate Hepatic Impairment (Panel A) | Severe Hepatic Impairment (Panel B)
Number analyzed (Participants) | 5 | 4
hours | 0.47 [0.47 to 0.53] | 0.50 [0.47 to 1.00]

6. Primary Outcome: Apparent Terminal Half-life (t1/2) of MK-3866
Description: Apparent t1/2 is the elimination half-life of MK-3866 from plasma.
Time Frame: Predose, 0.5 (end of infusion), 0.75, 1, 1.5, 2, 3, 4.5, 6, 8, 10, 12, 24, 48, and 72 hours postdose
Population: All treated participants with data available are included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Moderate Hepatic Impairment (Panel A) | Severe Hepatic Impairment (Panel B)
Number analyzed (Participants) | 5 | 4
hours | 6.54 (13.3) | 6.02 (4.16)

7. Primary Outcome: Clearance (CL) of MK-3866
Description: CL is the volume of plasma from which the study drug is completely removed per unit time.
Time Frame: Predose, 0.5 (end of infusion), 0.75, 1, 1.5, 2, 3, 4.5, 6, 8, 10, 12, 24, 48, and 72 hours postdose
Population: All treated participants with data available are included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hour
Arm/Group | Moderate Hepatic Impairment (Panel A) | Severe Hepatic Impairment (Panel B)
Number analyzed (Participants) | 5 | 4
Liters/hour | 4.16 (7.3) | 5.07 (41.3)

8. Primary Outcome: Volume of Distribution (Vz) of MK-3866
Description: Vz is the apparent volume of distribution during the terminal phase.
Time Frame: Predose, 0.5 (end of infusion), 0.75, 1, 1.5, 2, 3, 4.5, 6, 8, 10, 12, 24, 48, and 72 hours postdose
Population: All treated participants with data available are included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Moderate Hepatic Impairment (Panel A) | Severe Hepatic Impairment (Panel B)
Number analyzed (Participants) | 5 | 4
Liters | 39.3 (15.8) | 44.0 (27.4)

9. Secondary Outcome: Fraction of Dose of MK-3866 Excreted Unchanged in Urine (Fe)
Description: Fe is the amount of drug excreted unchanged in urine. Urine samples were collected in 4-hour intervals up to 24 hours post-dose. The study terminated prior to analysis of urine samples and therefore no data are available.
Time Frame: Predose, then pooled in the following increments: 0-4, 4-8, 8-12, 12-24 hours postdose
Population: Urine samples were collected but were not analyzed.
Arm/Group | Moderate Hepatic Impairment (Panel A) | Severe Hepatic Impairment (Panel B)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Renal Clearance (CLr) of MK-3866
Description: CLr is the volume of plasma from which the study drug is completely removed per unit time by the kidney (i.e., excreted into the urine). Urine samples are collected in 4-hour intervals up to 24 hours post-dose. The study terminated prior to analysis of urine samples and therefore no data are available.
Time Frame: Predose, then pooled in the following increments: 0-4, 4-8, 8-12, 12-24 hours postdose
Population: Urine samples were collected but were not analyzed.
Arm/Group | Moderate Hepatic Impairment (Panel A) | Severe Hepatic Impairment (Panel B)
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Number of Participants With at Least One Adverse Event (AE)
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to 14 days
Population: All treated participants are included.
Measure: Number; unit: Participants
Arm/Group | Moderate Hepatic Impairment (Panel A) | Severe Hepatic Impairment (Panel B)
Number analyzed (Participants) | 5 | 4
Participants | 2 | 1

12. Secondary Outcome: Number of Participants Who Discontinued the Study Due to an AE
Description: as for outcome 11
Time Frame: Up to 14 days
Population: All treated participants are included.
Measure: Number; unit: Participants
Arm/Group | Moderate Hepatic Impairment (Panel A) | Severe Hepatic Impairment (Panel B)
Number analyzed (Participants) | 5 | 4
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 14 days
Description: All treated participants are included.
Arm/Group | Moderate Hepatic Impairment (Panel A) | Severe Hepatic Impairment (Panel B)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 2/5 | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moderate Hepatic Impairment (Panel A) (N=5) | Severe Hepatic Impairment (Panel B) (N=4)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-06): https://cdn.clinicaltrials.gov/large-docs/66/NCT03295266/Prot_SAP_000.pdf